CLINICAL TRIAL: NCT06472089
Title: Multimodal Psychosocial Intervention for Caregivers of Patients Undergoing Hematopoietic Stem Cell Transplantation
Brief Title: BMT-CARE: Psychosocial Intervention for Transplant Caregivers
Acronym: BMT-CARE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, El-Jawahri, Areej,M.D., Associate Professor of Medicine, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 24-013
Record Dates: First submitted 2024-06-09; First posted 2024-06-24 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-10

CONDITIONS: Bone Marrow Transplant Complications; Hematologic Malignancy
Keywords: Neoplasms by Site; Hematologic Diseases; Neoplasms; Hematologic Neoplasms
MeSH Terms: conditions — Hematologic Neoplasms; Neoplasms by Site; Hematologic Diseases; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- BMT-CARE (Experimental): Participants randomized to BMT-CARE plus usual care will complete the following:
  * Questionnaires at baseline, and days 60, 90 and 180 post HCT.
  * Receive the BMT-CARE intervention from enrollment up to 60 days post-HCT. BMT-CARE is a -6-session caregiver-directed cognitive behavioral therapy (CBT)-based psychosocial intervention that integrates HCT-related education with CBT strategies to enhance caregiver knowledge and skills.
  * Receive usual care as per HCT practice which entails meeting a transplant social worker prior to HCT and as needed for extra visits.
  Interventions: Behavioral: BMT-CARE
- Usual Care (Active Comparator): Participants randomized to usual care will complete the following
  * Questionnaires at baseline, and days 60, 90 and 180 post HCT.
  * Receive usual care as per HCT practice which entails meeting a transplant social worker prior to HCT and as needed for extra visits.
  Interventions: Behavioral: Usual Care

INTERVENTIONS:
Behavioral: BMT-CARE — Therapist-delivered psychosocial intervention comprised of 6 sessions
  Arms: BMT-CARE
Behavioral: Usual Care — Meeting a transplant social worker prior to HCT and as needed for extra visits
  Arms: Usual Care

SUMMARY:
The goal of this study is to evaluate whether a psychological intervention (BMT-CARE) is effective at improving the quality of life in caregivers and patients treated with hematopoietic cell transplant compared to usual care, and to identify critical facilitators and barriers for BMT-CARE implementation and adoption.

DETAILED DESCRIPTION:
This is a randomized clinical trial to determine whether a psychosocial intervention (BMT-CARE) is effective at improving the quality of life and reducing psychosocial distress of caregivers and patients treated with hematopoietic cell transplant (HCT). The BMT-CARE intervention was developed with the goal of improving the experience and needs of caregivers of patients treated with HCT.

Caregivers will be randomized into one of the two study groups: BMT-CARE plus usual care, or usual care.

Participation in this study is expected to last up to 180 days after HCT.

Investigators expect that about 400 caregivers and up to 400 patients treated with HCT will take part in this research study.

The National Institutes of Health is supporting this research by providing funding.

ELIGIBILITY:
Caregiver Inclusion Criteria:

* Adult caregivers (≥18 years) relative or friend of a patient identified as living with them or having in-person contact with them at least twice a week.
* Caregiver of a patient receiving allogeneic or autologous HCT for the treatment of cancer.
* Ability to read and respond to survey questions in English, Spanish or with minimal assistance from an interpreter.

Caregiver Exclusion Criteria:

* Caregivers of patients undergoing HCT for a benign hematologic condition or undergoing outpatient HCT.
* Caregivers with a major untreated psychiatric or cognitive condition which the treating oncology clinicians believes interferes with the capacity to provide informed consent.
* Caregivers of patients who have already undergone HCT within the past 5 years

Patient Inclusion Criteria:

* Adult patients (≥18 years) with a hematologic malignancy and planned admission for autologous or allogeneic HCT.
* Ability to respond to questions in English, Spanish, or with minimal assistance from an interpreter.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2025-01-10 (Actual); Primary Completion 2028-05 (Estimated); Study Completion 2029-02 (Estimated)

PRIMARY OUTCOMES:
Caregiver quality of life (QOL) as measured by the Caregiver Oncology Quality of Life (CARGOQOL) questionnaire | Up to 60 days post-HCT
  Compare caregiver QOL as measured by the CARGOQOL between the two study groups. The CARGOQOL ranges from 0-100 with higher scores indicating better QOL

SECONDARY OUTCOMES:
Caregiver quality of life (QOL) as measured by the Caregiver Oncology Quality of Life (CARGOQOL) questionnaire | Up to 180 days post-HCT
  Compare caregiver QOL as measured by the CARGOQOL between the two study groups. The CARGOQOL ranges from 0-100 with higher scores indicating better QOL
Caregiving burden as measured by the Caregiver Reaction Assessment (CRA) questionnaire | Up to 180 days post-HCT
  Compare caregiving burden as measured by the CRA between the two study groups. The CRA ranges from 24-120 with higher scores indicating greater caregiving burden
Caregiver depression symptoms as measured by the Hospital Anxiety and Depression (HADS-Depression) Scale | Up to 180 days post-HCT
  Compare caregiver depression symptoms as measured by the HADS-Depression between the study groups. The HADS-Depression ranges from 0-21 with higher scores indicating worse depression symptoms
Caregiver anxiety symptoms as measured by the Hospital Anxiety and Depression (HADS-Anxiety) Scale | Up to 180 days post-HCT
  Compare caregiver anxiety symptoms as measured by the HADS-Anxiety between the study groups. The HADS-Anxiety ranges from 0-21 with higher scores indicating worse anxiety symptoms
Caregiver coping as measured by the Measure of Current Status-A (MOCS-A) questionnaire | Up to 180 days post HCT
  Compare caregiver coping as measured by the MOCS-A between the two study groups. The scale ranges from 0-52 with higher scores indicating higher coping skills
Caregiver self-efficacy as measured by the Cancer Self-Efficacy-transplant (CASE-t) questionnaire | Up to 180 days post-HCT
  Compare caregiver self-efficacy as measured by the CASE-t between the two study groups. The scale ranges from 0-170 with higher scores indicating better self-efficacy

OTHER OUTCOMES:
Patient quality of life as measured by the Functional Assessment of Cancer Therapy-BMT (FACT-BMT) questionnaire | Up to 180 days post-HCT
  Compare patient QOL as measured by the FACT-BMT between the two study groups. Score range 0-196 and higher scores indicate better QOL
Patient depression symptoms as measured by the Hospital Anxiety and Depression (HADS-Depression) scale | Up to 180 days post-HCT
  Compare patient depression symptoms as measured by the HADS-Depression between the study groups. The HADS-Depression ranges from 0-21 with higher scores indicating worse depression symptoms
Patient anxiety symptoms as measured by the Hospital Anxiety and Depression (HADS-Anxiety) scale | Up to 180 days post-HCT
  Compare patient anxiety symptoms as measured by the HADS-Anxiety between the study groups. The HADS-Anxiety ranges from 0-21 with higher scores indicating worse anxiety symptoms
Patient symptom burden as measured by the Revised Edmonton Symptom Assessment Scale -Revised (ESAS-r) | Up to 60 days post-HCT
  Compare patient symptom burden as measured by the ESAS-r between the study groups. Scor range 0-100 and higher scores indicate worse symptom burden.
Patient medication adherence as measured by the Medication Adherence Report Scale (MARS-5) | Up to 180 days post HCT
  Compare patient medication adherence as measured by the MARS-5 between study groups. Score range 5-25 with higher scors indicating better adherence.
Rate of caregiver healthcare utilization as self-reported by caregivers | At 180 days post HCT
  Compare Rates of caregiver healthcare utilization (e.g., hospitalizations, emergency department visits) between study groups.
Rate of caregiver adherence to primary care visits and age-appropriate cancer screening as self-reported by caregivers | At 180 days post HCT
  Compare rates of caregiver adherence to primary care visits and age-appropriate cancer screening between study groups
Rates of caregiver mental health resources utilization as self-reported by caregivers | At day 180 post HCT
  Compare rates of caregiver mental health resource utilization between study groups
Rate of patient healthcare utilization as self-reported by patients and extracted from the electronic medical record | At 180 days post HCT
  Compare rates of patient healthcare utilization (eg., hospitalizations, emergency department visits) between the study groups.
Rates of patient mental health resources utilization as self-reported by patients | At day 180 post HCT
  Compare rates of patient mental health resource utilization between study groups
Rates of acute and/or chronic graft-versus host disease based on data gathered from the electronic medical record | At day 180 post HCT
  Compare the rates of acute and/or chronic graft-versus-host disease between study groups

CONTACTS AND LOCATIONS:
Overall Officials: Areej El-Jawahri, MD, Principal Investigator — Massachusetts General Hospital; Jamie Jacobs, PhD, Principal Investigator — Massachusetts General Hospital
Locations (3):
- United States (3):
  - University of Alabama at Brimingham, Birmingham, Alabama
  - Moffitt Cancer Center, Tampa, Florida
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Partners Innovations team at http://www.partners.org/innovation